CLINICAL TRIAL: NCT00908518
Title: Postoperative Cognitive Dysfunction and Perioperative Myocardial Ischemia: Comparing Total IV Anesthesia and Inhalation Anesthesia.
Brief Title: The Difference in Postoperative Cognitive Dysfunction and Myocardial Ischemia Between Propofol and Isoflurane
Acronym: POCD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Ron Flaishon MD, Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC-08-RF-514-CTIL
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Cognitive Dysfunction; Cardiac Morbidity
Keywords: Cognitive dysfunction; Cardiac morbidity; anesthesia
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Total Intravenous Anesthesia: Propofol based anesthesia
- Inhaled anesthesia: Isoflurane based anesthesia

SUMMARY:
The progressive aging of the general population cause increase in number of extensive and long surgeries in older patients. Age is a risk factor for perioperative myocardial ischemia and Postoperative Cognitive Dysfunction (POCD) The suggested study will deal with the above-mentioned complication in patients older then 65 years undergoing major non-cardiac surgeries.

It has been shown that Isoflurane and sevoflurane may have a cardio-protective effect after cardiac surgery involving cardio-pulmonary bypass, and it was recommended that isoflurane should be used in these cases. A question was raised but haven't been answered yet, whether this cardio-protective effect exists also in non-cardiac major surgery.

The aim of this study is to evaluate whether there is a difference in the occurrence of postoperative cognitive dysfunction and perioperative myocardial ischemia between total intravenous anesthesia using propofol and isoflurane based anesthesia.

DETAILED DESCRIPTION:
The progressive aging of the general population cause increase in number of extensive and long surgeries in older patients. Age is a risk factor for perioperative myocardial ischemia and Postoperative Cognitive Dysfunction (POCD) The suggested study will deal with the above-mentioned complication in patients older then 65 years undergoing major non-cardiac surgeries.

It has been shown that Isoflurane and sevoflurane may have a cardio-protective effect after cardiac surgery involving cardio-pulmonary bypass, and it was recommended that isoflurane should be used in these cases. A question was raised but haven't been answered yet, whether this cardio-protective effect exists also in non-cardiac major surgery.

The aim of this study is to evaluate whether there is a difference in the occurrence of postoperative cognitive dysfunction and perioperative myocardial ischemia between total intravenous anesthesia using propofol and isoflurane based anesthesia.

The suggested study is a randomized controlled study. 500 patients older then 65 years undergoing elective non-cardiac major surgeries will be studied.

On the day prior to surgery the patient will take a series computerized cognitive tests (Mindstream® cognitive health assessment, neurotrax®, Modiin, Israel). At the holding area before entering the operating room (OR) the patients will be randomly assigned to one of two study groups.

Group 1 -IA: anesthesia will be maintained using Isoflurane carried by O2/air. Group 2 - TIVA : anesthesia will be maintained with propofol. The patients will be followed for 3 months post-operatively. Cognitive function will be assessed 7 days and 3 months postoperatively using computerized tests and telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Patients that refuse or unable to sign an informed consent

Exclusion Criteria:

* Patients with any unstable disease
* Patients treated with medication affecting the nervous system
* Patients with earring difficulty
* Patients that will not be able to participate in the study due to language barrier

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 500 patients older then 65 year, scheduled for elective non-cardiac, non-neuro surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
to evaluate whether there is a difference in the occurrence of POCD | 3 months

SECONDARY OUTCOMES:
To evaluate whether there is a difference in the occurrence of post-operative cardiac morbidity | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Ron Flaishon, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel